CLINICAL TRIAL: NCT00472238
Title: Effects of Endurance Training on Patients With Reduced LVEF and Cardiac Resynchronisation Therapy Especially for Cardiac Arrhythmias
Brief Title: Effects of Endurance Training on Patients With Reduced Left Ventricular Ejection Fraction (LVEF) and Cardiac Resynchronisation Therapy Especially for Cardiac Arrhythmias
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. Dirk Müller, Charité Campus Benjamin Franklin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBF-2007001; 001
Record Dates: First submitted 2007-05-10; First posted 2007-05-11 (Estimated); Last update posted 2008-11-20 (Estimated); Status verified 2007-05

CONDITIONS: Heart Failure; Cardiac Resynchronisation Therapy; Sudden Cardiac Death
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac | interventions — Endurance Training; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1, Training (Experimental): Group for training therapy
  Interventions: Behavioral: exercise training
- 2, Control (Active Comparator)
  Interventions: Behavioral: endurance training

INTERVENTIONS:
Behavioral: endurance training — control group.
  Arms: 2, Control
Behavioral: exercise training — Treadmill exercise training to optimize physical endurance
  Arms: 1, Training

SUMMARY:
A severely reduced left ventricular ejection fraction is associated with increased mortality due to pump failure as well as to malignant ventricular arrhythmia. We hypothesize that targeted training may lead to improved survival and to increased parameters of risk stratification for malignant arrhythmia. Additionally, the training may lead to an improved psychological and mental condition of the patients

ELIGIBILITY:
Inclusion Criteria:

* CRT Device

Exclusion Criteria:

* refused informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2007-08; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
left ventricular function | 3 months
aerobic threshold | 3 months

SECONDARY OUTCOMES:
quality of life | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Müller, MD, PhD, Principal Investigator — Charite University, Berlin, Germany; Fernando C Dimeo, MD, PhD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité campus Benjamin Franklin, Berlin, State of Berlin, Germany